CLINICAL TRIAL: NCT00419315
Title: Primary Care Based Disease Management for Alcohol Dependence
Brief Title: A Randomized Clinical Trial of Alcohol Care Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 06-058
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Alcohol Dependence
Keywords: alcoholism; primary care; treatment
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alcohol Care Management (Experimental): Care management for alcohol dependence delivered in primary care
  Interventions: Behavioral: Alcohol Care Management
- Usual Care (Active Comparator): Usual care included a referral to specialty addiction treatment
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Alcohol Care Management — Care management for alcohol dependence with a focus on pharmacotherapy
  Arms: Alcohol Care Management
Behavioral: Usual Care — Usual care included a referral to a specialty addiction treatment program.
  Arms: Usual Care

SUMMARY:
A randomized study of Alcohol Care Management for the treatment of alcohol dependence in primary care settings.

DETAILED DESCRIPTION:
Background: Alcohol dependence is one of the leading causes of disability worldwide. Despite the availability of efficacious treatments less than 20% of individuals with alcohol dependence are actively engaged in treatment. Within the VA system systematic screening was implemented to increase the identification of patients with both abuse and dependence. However, there continues to be a marked discrepancy in the care offered or accessed among those identified with alcohol dependence. Existing treatment guidelines suggest that all persons with dependence receive care in specialty addiction treatment. Data from our center indicate that among those individuals screened in primary care who have AUDIT - C scores of >7, only 30% are formally evaluated with 50% receiving only brief advice and 20% having no evidence of assessment or referral. Of those assessed and referred to specialty care only 60% attend an initial visit and only 33% meet the EPRP performance measure of 2 visits per month for 90 days. This disparity in treatment access exists even though Veterans self report a desire to cut down and readiness to change drinking behaviors. (VA ACQUIP) and a willingness to consider pharmacotherapy.

Aims: Available evidence suggests that primary care may be a key component in the identification of alcohol dependent patients, delivery of initial interventions, and to the success of addiction treatment. Indeed, the vast majority of screening and new case identification occurs within primary care. The primary aims of this proposal are to test the effectiveness of a primary care based Alcohol Care Management (ACM) program and to evaluate the barriers and facilitators to accessing and engaging individuals into treatment. The ACM program uses a Behavioral Health Specialist to deliver care focused on the use of pharmacotherapy in combination with psychosocial support (Medication Management). This model may overcome barriers to care such as frequent intensive visit schedules often required in specialty settings, stigma associated with specialty care or group therapy approaches, access to specialty care in remote areas, and the current focus on a 12 step model of treatment. Secondary aims are to establish the acceptability of primary care based treatments and defining treatment modifiers such as age, barriers, co-occurring depression, and pharmacogenetic response.

ELIGIBILITY:
Inclusion Criteria:

* be men and women = 18 years of age;
* meet criteria for alcohol dependence;
* drink more than an average of 2 drinks per day prior to study entry (over the last 60 days);
* have adequate hearing to participate in assessment

Exclusion Criteria:

* show no evidence of current abuse or dependence of illicit substances other than marijuana;
* no current hallucinations;
* no current symptoms of mania;
* be relatively cognitively intact
* not actively participate in specialized addition or behavioral health treatment within the prior 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Oslin DW, Lynch KG, Maisto SA, Lantinga LJ, McKay JR, Possemato K, Ingram E, Wierzbicki M. A randomized clinical trial of alcohol care management delivered in Department of Veterans Affairs primary care clinics versus specialty addiction treatment. J Gen Intern Med. 2014 Jan;29(1):162-8. doi: 10.1007/s11606-013-2625-8. Epub 2013 Sep 20. PMID 24052453
- [Derived] Rotenberg JR, Leong SH, Maisto SA, McKay JR, Possemato K, Ingram E, Oslin DW. Post-intervention Durability of Alcohol Care Management: 1-Year Follow-up of a Randomized Controlled Trial. J Gen Intern Med. 2018 Oct;33(10):1626-1628. doi: 10.1007/s11606-018-4567-7. No abstract available. PMID 30003479

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Care management for alcohol dependence
  Alcohol Care Management: Care management for alcohol dependence with a focus on pharmacotherapy
- Arm 2: Usual care
  Alcohol Care Management: Care management for alcohol dependence with a focus on pharmacotherapy
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 85 | 78
Completed | 85 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 85 | 78 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.4) | 57.1 (10.1) | 56 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 85 | 73 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 44 | 94
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 78 | 163
% Days of Heavy Drinking [Mean (Standard Deviation); unit: % days of heavy drinking] — The measures the percent of days in the 60 days prior to randomization in which a participant drank more than 4 standard drinks (3 or more for women) in a given day.
  % days of heavy drinking | 54.5 (53.8) | 54.7 (33.6) | 54.6 (44.1)
The number of Subjects Engaged in Treatment at Baseline [Number; unit: Participants engaged in treatment] — This was a measure of the proportion of patients engaged in addiction treatment at the time of randomization. It was a requirement that no of the subjects were engaged at baseline.
  Participants engaged in treatment | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Engagement
Description: This measured the percentage of subjects who attended at least 2 clinical addiction sessions in a given month. The outcome presented is the percentage during the 6th month of the trial.
Time Frame: 6 months
Measure: Number; unit: percentage of participants engaged
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 85 | 78
percentage of participants engaged | 36 | 9

2. Secondary Outcome: Percent Days of Heavy Alcohol Use
Description: This is a measure during the 6 month of the percentage of 30 days in which a subject had at least 1 day of heavy drinking as defined by drinking more than 4 standard drinks in a day (3 or more for women).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 73 | 67
percentage of heavy drinking days | 18.0 (30.7) | 25.6 (33.0)

ADVERSE EVENTS:
Time Frame: the 6 months of the intervention trial
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/78
Other Adverse Events (participants affected / at risk) | 0/85 | 0/78

LIMITATIONS AND CAVEATS:
The data presented in the results does not provide a true measure of the longitudinal effects done with GEE modeling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No